CLINICAL TRIAL: NCT05775042
Title: A Phase II Clinical Study Evaluating the Efficacy and Safety of CM338 Injection in Subjects With Immunoglobulin A Nephropathy
Brief Title: Clinical Study of CM338 in the Treatment of Immunoglobulin A Nephropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM338-105101
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): CM338 will be injected subcutaneously.
  Interventions: Biological: CM338
- Group B (Experimental): CM338 will be injected subcutaneously.
  Interventions: Biological: CM338
- Group C (Experimental): CM338 will be injected subcutaneously.
  Interventions: Biological: CM338

INTERVENTIONS:
Biological: CM338 — CM338 injection

SUMMARY:
This study is a multicenter, randomized phase II clinical study to evaluate Efficacy and safety, while observing pharmacokinetic profiles, pharmacodynamic effects, and immunogenicity of CM338 in subjects with Immunoglobulin A(IgA) nephropathy.

DETAILED DESCRIPTION:
In 1968, immunoglobulin A nephropathy (IgAN) was developed by French pathologist Dr. Jean Berger and his colleague Dr. Nicole Hinglais that what is described as glomerular "immunoglobulin A (IgA)-immune globule" - immune globule Protein G (IgG) intercapillary deposition" of kidney disease, the main pathological feature of which is on the glomerulus IgA deposition, usually accompanied by local cell proliferation and stromal dilation. Since there is not enough specificity and spirit Biomarkers of sensitivity, the only way to confirm the diagnosis is renal biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-75.
* Understand the nature of the study and sign the Informed Consent Form voluntarily.
* Take effective contraception measures throughout the study period.

Exclusion Criteria:

* Used other investigational drugs within 30 days before the first study administration.
* With previous history of Human immunodeficiency virus(HIV) infection.
* Treponema pallidum antibody positive in screening period.
* May have active Mycobacterium tuberculosis infection.
* Major surgery is planned during the study.
* Other reasons the investigator believes that the subject is not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events of CM338 in subjects with immunoglobulin A nephropathy | up to week 112
  To evaluate the incidence of adverse events, including abnormalities of laboratory examination, physical examination, vital signs, 12-lead electrocardiogram (12-ECG) and others.

CONTACTS AND LOCATIONS:
Overall Officials: Jicheng Lv, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639